CLINICAL TRIAL: NCT06049667
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics and Preliminary Efficacy of NTQ2494 Tablets in Patients With Advanced Hematological Malignancies
Brief Title: A Phase 1 Clinical Trail of NTQ2494 Tablets in Patients With Advanced Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTQ2494-23101
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NTQ2494 (Experimental): For each dose level, multiple doses of NTQ2494 tablets will be administered as 28-day treatment (per cycle).
  Interventions: Drug: NTQ2494 tablet

INTERVENTIONS:
Drug: NTQ2494 tablet — Drug: NTQ2494 tablet Part 1: Dose escalation, single and multiple doses of NTQ2494 with dose modifications based on tolerability criteria.
  For each dose level, a single dose of NTQ2494 tablets will be first administered orally, then continuous 28-day treatment will start (per cycle).
  Part 2: Dose expansion, recommended doses from Part 1. For each dose level, multiple doses of NTQ2494 tablets will be administered as 28-day treatment (per cycle).

SUMMARY:
NTQ2494 tablet, an anti-tumor molecular targeted drug, is an AXL kinase inhibitor.

The objectives were to evaluate the safety and tolerability, PK characteristics and preliminary efficacy of NTQ2494 tablets in patients with advanced hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years in age, male or female.
2. Relapsed/refractory AML patients.
3. ECOG performance status score is 0 to 2.
4. Life expectancy of at least 3 months.
5. Adequate bone marrow and good organ function.
6. Ability to understand the purpose and risks of the study and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Receiving anticancer therapy including immunotherapy, targeted therapy, endocrine therapy, radiotherapy and chemotherapy within 2 weeks or 5 half-lives (whichever is longer) prior to starting study treatment.
2. Receiving any other investigational agents within 4 weeks prior to starting study treatment.
3. Having major surgery within 4 weeks prior to starting study treatment, or intended to undergo surgery during the trail.
4. AML with any of the following: 1) acute promyelocytic leukemia; 2) AML with blast crisis of chronic myelogenous leukemia; 3) central nervous system leukemia.
5. Prior or current other malignancy (except cured noninvasive basal cell or squamous cell skin cancer and/or other cured carcinoma in situ; except for other malignancies that have achieved clinical cure for > 5 years and have not recurred within 5 years).History of severe cardiovascular or cerebrovascular disease.
6. Use of strong inhibitors or strong inducers of CYP3A4 or P-gp within 7 days prior to starting study treatment.
7. Receiving (attenuated) live vaccines within 4 weeks prior to starting study treatment and/or planning to receive (attenuated) live vaccines during the trial.
8. With unresolved clinically significant non-hematological toxicities from prior AML therapy (chemotherapy, targeted therapy, immunotherapy, radiotherapy and surgery), defined as any grade 2 or higher grade (CTCAE v5.0), alopecia and other events that are tolerable as judged by the investigator.
9. Patients who have received previous allogeneic hematopoietic stem cell transplantation; or received autologous hematopoietic stem cell transplantation within 3 months prior to starting study treatment.
10. Unable to swallow oral tablets, or other conditions seriously affecting gastrointestinal absorption judged by the investigator.
11. Patients with uncontrolled infections unsuitable for the trail judged by the investigator.
12. Known infection with hepatitis B, hepatitis C, HIV or Syphilis.
13. Known alcohol or drug dependence.
14. Patients with mental disorders or poor compliance.
15. Patients with a previous history of severe allergy to any drug or food.
16. Lactating or pregnant female, and females or males (or partners) who plan to pregnant and do not agree to use adequate contraception for the duration of the trail and up to 3 months after completion of the last study treatment.
17. Other reasons judged by the investigator that the patients unsuitable for the trail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerance dose (MTD) and dose limiting toxicity (DLT) | 30 days
  MTD is defined as the maximum dose level at which no more than 1 of 3 participants experience a DLT within the days of single dose and the first 28 days of multiple doses in dose escalation part.

SECONDARY OUTCOMES:
Cmax of single dose | At the end of Cycle 1 (each cycle is 28 days)
AUC0-t of single dose | At the end of Cycle 1 (each cycle is 28 days)
AUC0-∞ of single dose | At the end of Cycle 1 (each cycle is 28 days)
Tmax of single dose | At the end of Cycle 1 (each cycle is 28 days)
t1/2z of single dose | At the end of Cycle 1 (each cycle is 28 days)
Vz/F of single dose | At the end of Cycle 1 (each cycle is 28 days)
CLz/F of single dose | At the end of Cycle 1 (each cycle is 28 days)
λz of single dose | At the end of Cycle 1 (each cycle is 28 days)
MRT0-t of single dose | At the end of Cycle 1 (each cycle is 28 days)
Rac of AUC and Cmax of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
DF of AUC and Cmax of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
Css,max of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
Css,min of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
AUCss of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
Cav of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
Tss,max of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
t1/2 of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
Vz/F of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
  、Vz/F、CLss/F、λz of first 28 days of multiple doses.
CLss/F of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
λz of first 28 days of multiple doses | At the end of Cycle 1 (each cycle is 28 days)
Objective response rate (ORR) | through study completion, an average of 1 year
  ORR is defined as the proportion of subjects with confirmed CRc or PR.
Composite response (CRc) rate | through study completion, an average of 1 year
  CRc rate is defined as the proportion of subjects with confirmed CR or CRi or CRh.
Duration of response (DOR) | through study completion, an average of 1 year
  DOR is defined as the duration from the date of the first documented response of CR or PR to the date of the first documented recurrence or death.
Recurrence-free survival (RFS) | through study completion, an average of 1 year
  RFS is defined as the duration from the date of the first documented response of CRc to the date of the first documented recurrence or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China